CLINICAL TRIAL: NCT05220813
Title: Does Ilioinguinal Block Provide Satisfactory Analgesia During Transcatheter Aortic Valve Implantation Procedure? A Comparative Study
Brief Title: Ilioinguinal Nerve Block in Transcatheter Aortic Valve Implantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ismail Mohammed, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R 187/2021
Record Dates: First submitted 2022-01-22; First posted 2022-02-02 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local anesthetic group (control group) (Active Comparator): 44 patients will receive local infiltration anesthesia.
  Interventions: Drug: Lidocaine
- ilioinguinal iliohypogastric group (Active Comparator): 44patients will receive ilioinguinal iliohypogastric nerve blocks
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Lidocaine — local infiltration by lidocaine in the surgical site
  Arms: local anesthetic group (control group)
Drug: Bupivacain — 44patients will receive bupivacaine in ilioinguinal & iliohypogastric nerve blocks
  Arms: ilioinguinal iliohypogastric group

SUMMARY:
To assess the effect of iliohypogastric and ilioinguinal nerve block on the hemodynamic stability ,narcotic consumption and the rate of conversion to general anesthesia in patients undergoing transfemoral transcatheter aortic valve implantation (TF-TAVI).

ELIGIBILITY:
Inclusion Criteria:

* • Patients undergoing TF-TAVI.

  * Both sexes.
  * Age 18 and above

Exclusion Criteria:

* • Inability to tolerate supine position as in patients with musculoskeletal disease or back pain, OR in patients with congestive heart failure or with obstructive sleep apnea.

  * Patients with severe pulmonary hypertension (PAP>60 mmhg)
  * Barrier to communications as language barrier or dementia.
  * Patients' preference of general anesthesia.
  * Surgical consideration as transapical, subclavian approach, extensive TEE requirements.
  * Patients with history of allergy to any drugs used.
  * Patients with psychiatric disease.
  * Patients with neurocognitive or neurodegenerative disease.
  * Secondary exclusion criteria include abortion of the procedure, perioperative emergency conversion to general anesthesia and the need to cardiopulmonary resuscitation so the primary endpoint couldn't be detected in these conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
conversion to general anesthesia. | during the procedure (intraoperatively)
  Conversion to general anesthesia in other than procedure related causes.

SECONDARY OUTCOMES:
propofol dose | during the procedure (intraoperatively)
  Total dose of propofol per hour (0.025-0.075 mg /kg/min)
fentanyl dose | during the procedure (intraoperatively)
  total dose of fentanyl 1-2 microgram / kg
sedation score | during the procedure (intraoperatively)
  sedation score intraoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ismail Mohammed Ibrahim, Cairo, Egypt